CLINICAL TRIAL: NCT02668042
Title: Living Tissue Engineering Skin Substitutes Safety and Efficacy Studies for the Treatment of Difficult to Heal Wounds
Brief Title: The Activity of Tissue Engineering Skin Substitutes
Acronym: MSCs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xiaobing Fu, Academican, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHIH-PLAGH-ST-006
Record Dates: First submitted 2016-01-21; First posted 2016-01-29 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Difficult to Heal Wounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- liveness tissue skin (Experimental)
  Interventions: Biological: liveness tissue skin

INTERVENTIONS:
Biological: liveness tissue skin — liveness tissue skin safety and effectiveness for the treatment of difficult to heal wounds

SUMMARY:
The main purpose of this experiment was to evaluate the activity of tissue engineering skin substitutes safety and efficacy studies for the treatment of difficult to heal wounds

DETAILED DESCRIPTION:
This study for 6 months for a single center, open, randomized, controlled clinical trials before and after itself, test contains preliminary screening, treatment and follow-up after discharge of the patient.After treatment in patients with early debridement, in the case of no infection of living tissue engineering skin substitute transplantation, observe the wound healing after transplantation, chronic wound evaluation activity of tissue engineering skin substitutes in the efficacy and safety of wound healing after transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Meet difficult had 1 month or more to heal the wound patients
2. Who signed the informed consent of men or women older than 17 (pregnancy)
3. Has the ability to care for, has the ability to self signed informed consent, 7 to 17 years old must be signed by the guardian informed consent
4. The process of mental stability, can finish the test

Exclusion Criteria:

1. Known allergic to bovine collagen or gao min physique
2. the wound is greater than the10cm×10cm
3. People with mental illness, drug abusers and or other items
4. Pregnant women,Prepare a pregnancy or breast feeding women
5. 3 months participated in other similar experiment
6. Serious infectious disease not controller
7. With surgery, such as severe trauma stress situation
8. Can not meet the requirement of the long-term follow-up of patients

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Frequency of Adverse Events | 6 months
  Frequency and severity of Adverse Events

SECONDARY OUTCOMES:
Relative Wound Area Regression of 40% or More at 6 Week | 6 week

OTHER OUTCOMES:
Reduced pain | 6 months after treatment
  Reduced pain, measured by VAS scale and use of analgesics

CONTACTS AND LOCATIONS:
Overall Officials: xiaobing Fu, Principal Investigator — Chinese PLA General Hospital